CLINICAL TRIAL: NCT01303809
Title: Enhanced Recovery After Laparoscopic Sleeve Gastrectomy - a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Auckland Medical Research Foundation (Other)
Responsible Party: Principal Investigator, SACS, Professor Andrew G. Hill, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BariatricFastTrack
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Morbid Obesity
Keywords: Perioperative care; Fast-track; Enhanced Recovery After Surgery; ERAS; Obesity; Bariatric surgery; Laparoscopic Sleeve Gastrectomy
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERAS (Active Comparator): The perioperative management of the patients in this arm will be according to a fast-track protocol designed by the investigators. The preoperative component of this program is the same as routine practice. Intraoperative and postoperative components which are different to routine practice are as described in the intervention section. This protocol is based on current literature regarding Enhanced Recovery After Surgery (ERAS).
  Interventions: Other: Enhanced Recovery After Surgey for Sleeve Gastrectomy
- non ERAS (No Intervention): The perioperative management of patients in this arm will be according to routine practice currently implemented at our institution.

INTERVENTIONS:
Other: Enhanced Recovery After Surgey for Sleeve Gastrectomy — Intraoperative:
  1. Pre-op carbohydrate loading
  2. No pre-op GIK while NBM
  3. Pre-medication
  4. Dexamethasone 4mg as antiemetic, IV Paracetamol (first dose) Parecoxib 40mg
  5. Ondansetron regularly for first 48 hours and Cyclizine, Droperidol or Scopaderm as rescue antiemetics
  6. Fluid restriction
  7. Standardised method of anaesthesia
  8. Give 40ml 0.5% bupivacaine with adrenaline administered prior to placement of laparoscopic port sites
  9. 10ml 0.75% ropivacaine diluted to 50ml with 0.9% normal saline solution administered to surgical site prior to procedure
  Postoperative:
  1. Rescue PCA for up to 12 hours. Oxynorm 5mg for rescue pain. Oxycontin 20mg bd/prn postoperatively
  2. Maintenance IV fluids (60ml/hr plasmalyte to be stopped 0800 day 1 post op). Clear oral fluids 2 hours post op. Bariatric free oral fluids morning of day 1
  3. Post operative oxygenation
  4. Incentive spirometry
  5. Drains (e.g. IDC) removed in recovery
  6. Full mobilisation 4-8 hours post op)
  7. Early Follow up
  Other Names: ERAS for sleeve gastrectomy; Fast-Track for sleeve gastrectomy
  Arms: ERAS

SUMMARY:
The investigators wish to standardise and optimise perioperative care for consecutive patients undergoing laparoscopic sleeve gastrectomy for weight loss. The investigators will compare patients under a standardised perioperative care program to patients who undergo routine perioperative in our hospital and determine whether patients who had optimised perioperative care went home earlier and had fewer complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparascopic sleeve gastrectomy for weight loss by surgeons who have agreed to participate in the study
* Surgery occurs at Manukau Surgery Centre

Exclusion Criteria:

* Surgery not occuring in Manukau Superclinic

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | day of discharge
  The trial intends to investigate whether median length of hospital stay for patients under a standardised optimised perioperative care program is less than patients who have routine perioperative care that undergo the same operation.

SECONDARY OUTCOMES:
Complications | 30 days
  The study will investigate complication rate for each group identifying incidence, type and severity of complication according to the Clavien Dindo Classification system
Readmission rates | 30 days
  The number of patients per group who represent to hospital for any reason during a 30 day period after the day of surgery
Postoperative fatigue | Baseline and postoperative days 1, 7 and 14
  A measure functional recovery after surgery as measured by the validated surgical recovery scale.
Compliance to the ERAS protocol | through to day 1 postoperatively
  Prospectively recording whether components of the ERAS programme are being carried out as per protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Manukau Surgery Centre, Auckland, New Zealand

REFERENCES:
- [Derived] Lemanu DP, Singh PP, Berridge K, Burr M, Birch C, Babor R, MacCormick AD, Arroll B, Hill AG. Randomized clinical trial of enhanced recovery versus standard care after laparoscopic sleeve gastrectomy. Br J Surg. 2013 Mar;100(4):482-9. doi: 10.1002/bjs.9026. Epub 2013 Jan 21. PMID 23339040